CLINICAL TRIAL: NCT01441427
Title: Enteral Granulocyte Colony Stimulating Factor and Erythropoietin Early in Life Increases Feeding Tolerance in Preterm Infants: A Randomized Controlled Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU 548/2010
Record Dates: First submitted 2011-09-18; First posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Feeding Intolerance; Necrotizing Enterocolitis
Keywords: feeding intolerance; recombinant growth factors; G-CSF; EPO; necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- G-CSF (Experimental)
  Interventions: Drug: rh G-CSF
- EPO (Experimental)
  Interventions: Drug: rh EPO
- G-CSF and EPO (Experimental)
  Interventions: Drug: recombinant human G-CSF, and rhEPO; Drug: rh G-GSF and rh EPO together
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human G-CSF, and rhEPO — G-CSF 4.5 microgram /kg/day enteral EPO 88 mIU/kg/day enteral
  Arms: G-CSF and EPO
Drug: rh G-CSF — Dosage: 4.5 µg/ kg (diluted into 1 ml distilled water) administered once daily by an orogastric tube till the enteral intake reached 100 mL/kg of milk, or after a maximum of seven days.
  Arms: G-CSF
Drug: rh EPO — Dosage: 88 IU/ kg once daily (diluted into 1 ml distilled water) administered by an orogastric tube till the enteral intake reached 100 mL/kg of milk, or after a maximum of seven days.
  Arms: EPO
Drug: rh G-GSF and rh EPO together — EPO dosage: 88 IU/ kg once daily i.e 88000 mU/kg/day (diluted into 1 ml distilled water) administered by an orogastric tube till the enteral intake reached 100 mL/kg of milk, or after a maximum of seven days.G-CSF dosage: 4.5 µg/ kg (diluted into 1 ml distilled water) administered once daily by an orogastric tube till the enteral intake reached 100 mL/kg of milk, or after a maximum of seven days.
  Arms: G-CSF and EPO
Drug: Placebo — distilled water :1 ml distilled water administered by an orogastric tube till the enteral intake reached 100 mL/kg of milk, or after a maximum of seven days.
  Arms: Placebo

SUMMARY:
With preterm birth, the ingestion of amniotic fluid containing enterocyte trophic factors ceases abruptly. This likely predisposes them to villous atrophy feeding intolerance and necrotizing enterocolitis(NEC) once feedings are instituted.Granulocyte Colony-Stimulating Factor (G-CSF) and Erythropoietin (EPO) have important non-hematopoietic roles in human developmental biology. Among these roles, they have trophic actions on villous height and bowel length of the developing intestine.The aim of this study is to evaluate the efficacy of enteral recombinant human G-CSF and recombinant human EPO in prevention of feeding intolerance and /or NEC in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* premature neonates < 33 weeks gestational age

Exclusion Criteria:

* major congenital anomalies
* prior use of cytokines

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The times taken to establish quarter, half, three quarters, and full enteral feeding after the drug treatment (at least 150ml/kg/day). | one month
Time to stop parentral nutrition | one month
Day of onset of weight gain | one month
Duration of hospitalization | 2 months

SECONDARY OUTCOMES:
Necrotizing enterocolitis (NEC)stage (if any) | 2 months
  Bell and colleagues proposed a clinical staging system for NEC: infants with suspected NEC (stage I), definite NEC (stage II), or advanced NEC (stage III) (Bell et al., 1978).

REFERENCES:
- [Derived] El-Ganzoury MM, Awad HA, El-Farrash RA, El-Gammasy TM, Ismail EA, Mohamed HE, Suliman SM. Enteral granulocyte-colony stimulating factor and erythropoietin early in life improves feeding tolerance in preterm infants: a randomized controlled trial. J Pediatr. 2014 Dec;165(6):1140-1145.e1. doi: 10.1016/j.jpeds.2014.07.034. Epub 2014 Aug 23. PMID 25155966